CLINICAL TRIAL: NCT03640559
Title: Multicenter, Double-blind, Placebo-controlled, Randomized, Parallel-group Study of Safety and Tolerability of Seroguard, Solution (JSC Pharmasyntez, Russia) in Patients Undergoing a Planned Laparoscopic Cholecystectomy
Brief Title: Safety and Tolerability of Seroguard Use
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmasyntez (Industry)
Collaborators: Sciencefiles (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SG -1/1014
Record Dates: First submitted 2018-08-16; First posted 2018-08-21 (Actual); Results first posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2018-08

CONDITIONS: Adhesion
Keywords: Adhesion; Safety
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Intervention Model Description: laparoscopic cholecystectomy
Who Masked: Participant, Investigator
Masking Description: The present study was planned as double-blind, placebo-controlled study. With the aim of maximum objectification of end point, neither Medical Investigator, nor patients had access to the code of healthcare institution.
  The test drug or the placebo were received by the sites as ready for use and blinded vials, 200 mL each. Each vial had individual number and identification of contents ("Drug A" or "Drug B"). Conformity of identification of Seroguard or the placebo was not disclosed to the sites.
  Before surgery, the Medical Investigator prepared required number of vials according to identification of the drug on the vial and identification of the group in randomization envelope of patient. Individual number of each vial administered to a patient was recorded in documentation of site.
Oversight: FDA-regulated Drug: No

ARMS (2):
- Placebo (Placebo Comparator): the group were having the administration of Placebo (saline 2.4 mL/kg IP)
  Interventions: Drug: Placebos
- Seroguard (Experimental): the group were having the administration of Seroguard 0.41 g/L solution, 2.4 mL/kg IP
  Interventions: Drug: Seroguard

INTERVENTIONS:
Drug: Seroguard
  Arms: Seroguard
Drug: Placebos
  Arms: Placebo

SUMMARY:
The performed study of safety and tolerability of Seroguard, solution (JSC Pharmasyntez, Russia) in patients, undergoing planned laparoscopic cholecystectomy, demonstrated that patients from the both groups had the similar safety profile

DETAILED DESCRIPTION:
The present study was conducted as multicenter, randomized, double-blind, parallel group clinical study. After successful completion of screening procedures, patient underwent a planned laparoscopy. Randomization of patients into groups was performed on the day of surgery using envelops. The test drug or the placebo were used at the completion stage of surgery. Monitoring of patient on inpatient basis was performed for 6 days after completion of surgery. Discharge of patient from the hospital with no contraindications was possible on Day 7 of the study. In this case the follow-up of patient was performed on outpatient basis. Follow-up was performed for 4 weeks before Day 28 of the study. Study procedures aimed at evaluation of safety and tolerability of using the test drug or the placebo were identical in main and control groups.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients.
2. Age from 18 to 75 years, inclusive.
3. Signed informed consent form.
4. One of the following diagnoses as per International classification of diseases -10:

   4.1. K80.1 Calculus of gallbladder with other cholecystitis 4.2. K80.2 Calculus of gallbladder without cholecystitis
5. Indications for planned laparoscopic cholecystectomy.

Exclusion Criteria:

1. Recall of informed consent by patient.
2. Non-compliance with the rules of participating in the study by patient.
3. Getting pregnant.
4. Required conversion during surgery.
5. Required repeated surgery.
6. Development of diseases described in non-inclusion criteria, required use of drugs not provided by the protocol in patient.
7. Another reasons appeared during the study and interfering conduction of the study as per the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-05-19 (Actual); Primary Completion 2015-10-04 (Actual); Study Completion 2015-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Shurygin, PhD, Study Director — Pharmasyntez

REFERENCES:
- [Background] The Federal Law dated 12.04.2010 №61-ФЗ "On drug circulation" (as amended Federal Laws dated 27.07.2010 N 192-ФЗ, dated 11.10.2010 N 271-ФЗ, dated 29.11.2010 N 313-ФЗ, dated 06.12.2011 N 409-ФЗ, dated 25.06.2012 N 93-ФЗ, dated 25.12.2012 N 262-ФЗ, dated 02.07.2013 N 185-ФЗ, dated 25.11.2013 N 317-ФЗ, dated 12.03.2014 N 33-ФЗ, dated 22.10.2014 N 313-ФЗ)
- [Background] The Order of the Ministry of Health, the Russian Federation, No 266 dated 19.06.2003.
- [Background] GOST R 52379-2005 "National standard of the Russian Federation "Good Clinical Practice" (approved by the Order of the Federal Agency for Technical Regulation and Metrology dated 27th of September, 2005 No 232-ст).
- [Background] Declaration of Helsinki, World Medical Association (as revised, approved at 64th General Assembly, Fortaleza (Brazil, 2013))
- [Background] Guideline on inspection of medicinal drugs. Volume I. Grif and K, 2013. - 328 p.
- [Background] Bonferroni, C. E. (1936). Teoria statistica delle classi e calcolo delle probabilità, Pubblicazioni del R Istituto Superiore di Scienze Economiche e Commerciali di Firenze.
- [Background] Stata Statistical Software: Release 13. College Station T:SL, 2.

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: the group were having the administration of Placebo (saline 2.4 mL/kg IP)
  Placebos
- Seroguard: the group were having the administration of Seroguard 0.41 g/L solution, 2.4 mL/kg IP
  Seroguard
Period: Overall Study
Arm/Group | Placebo | Seroguard
Started | 25 | 25
Completed | 23 | 24
Not Completed | 2 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Seroguard | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 20 | 39
  >=65 years | 4 | 4 | 8
Age, Continuous [Mean (Full Range); unit: years] | 49.3 [22 to 68] | 51.5 [22 to 66] | 50.4 [22 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  Russia | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Evaluation of safety of the study drugs Seroguard and the Placebo will be performed for all the study subjects at Visits 1-11, based on account of parameter:
  * Vital signs (body temperature, BP, HR, RR)
  * Laboratory investigations:
  * Blood chemistry - total protein, glucose, ALT, AST, total bilirubin, alkaline phosphatase, amylase, creatinine
  * Complete blood count - RBC, WBC, platelet count, hemoglobin, hematocrit, WBC differential, ESR
  * Coagulogram - coagulation time, international normalized ratio (INR), thrombin time, activated partial thromboplastin time (APTT)
  * Urinalysis - color, transparency, pH, specific gravity, protein, glucose, WBC, RBC, bacteria, casts, salts
  * 12-channel ECG data - heart rate [HR], PR, QRS, QT intervals and calculated QTc interval
  * USG data
  * Incidence of adverse reactions
  * Incidence of serious adverse reactions
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Seroguard
Number analyzed (Participants) | 23 | 24
Participants | 16 | 17

ADVERSE EVENTS:
Arm/Group | Placebo | Seroguard
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/23 | 2/24
Other Adverse Events (participants affected / at risk) | 16/23 | 17/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=23) | Seroguard (N=24)
pains in the right supraclavicular area (Surgical and medical procedures) | 0 (0) | 1 (1)
Leukocytosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Increased blood pressure up to 220/100 mm (Cardiac disorders) | 0 (0) | 1 (1)
Misbirth (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=23) | Seroguard (N=24)
Hyperthermia (Surgical and medical procedures) | 11 (24) | 12 (18)
Headache (General disorders) | 6 (9) | 5 (16)
Arterial hypertension (Cardiac disorders) | 1 (1) | 3 (7)
Pain in lower extremities (General disorders) | 1 (1) | 2 (2)
Back pain (Nervous system disorders) | 0 (0) | 1 (2)
Pain in the right hypochondrium (Hepatobiliary disorders) | 7 (10) | 3 (9)
Sore throat (Infections and infestations) | 0 (0) | 3 (3)
Pain in right side of chest (Surgical and medical procedures) | 2 (2) | 0 (0)
Epigastric pain (Gastrointestinal disorders) | 5 (7) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (3) | 1 (3)
Pain in postoperative wound (Surgical and medical procedures) | 3 (3) | 0 (0)
Kidney pain (Renal and urinary disorders) | 1 (2) | 0 (0)
Pain in the right infraclavicular region (Surgical and medical procedures) | 3 (3) | 1 (1)
Hypertensive crisis (Cardiac disorders) | 0 (0) | 2 (2)
Dizziness (General disorders) | 1 (1) | 3 (4)
Constipation (Gastrointestinal disorders) | 3 (6) | 2 (3)
Toothache (General disorders) | 0 (0) | 1 (2)
Burning sensation (General disorders) | 0 (0) | 3 (8)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (2)
Cholemesis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Palpitation (Cardiac disorders) | 0 (0) | 1 (2)
Weakness (General disorders) | 1 (2) | 3 (5)
Nausea (Gastrointestinal disorders) | 2 (3) | 3 (3)
Heaviness in epigastrium (Gastrointestinal disorders) | 3 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No